CLINICAL TRIAL: NCT04777305
Title: The POWER BARIATRIC Trial: Physical Outcomes With Exercise Regimens on BARIATRIC Patients
Acronym: POWER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel Aviv University (Other)
Collaborators: Herzliya Medical Center (Other)
Responsible Party: Principal Investigator, Gepner Yftach, Dr. Gepner Yftach, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0010-20-HMC
Record Dates: First submitted 2021-02-08; First posted 2021-03-02 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Obesity; Muscle Loss; Adiposity
Keywords: Obesity; Bariatric Surgery; Muscle mass loss; exercise training
MeSH Terms: conditions — Obesity; Muscular Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic exercise training (Experimental): The aerobic exercise training group, weeks 5-8 after surgery: this training will consist of 30 min. of walking, 3 times per week at an intensity of 60-70% of peak VO2 or RPE 6-7 on the Borg scale.
  Weeks 9-26 after surgery: this training will consist of 60 minutes of exercise, 3 times per week at an intensity of 65-80% of peak VO2 or RPE 6-8 on the Borg scale. The aerobic exercises will consist of a treadmill or outside walking or running, stationary cycling or elliptical trainer in continuous and interval training.
  Interventions: Other: Physical activity training
- Resistance exercise training (Experimental): Resistance exercise training group, weeks 5-8 after surgery: this training will consist of 5-10 minutes of warmup, followed by 6-8 multi-joint exercises for major muscle groups, comprising 2 sets of 10 to 25 repetitions at 40% of the one-repetition maximum (1-RM) for each exercise. The intensity will increase on weeks 9-26 after surgery to 8-10 multi-joint exercises of 3-4 sets of 10 to 25 repetitions. For this training participants will use free-weights and body weight exercises.
  Interventions: Other: Physical activity training
- Combination exercise training (Experimental): The combination exercise training will consist of a combined aerobic and resistance exercise training sessions three times weekly. At weeks 5-8 after surgery the sessions will include 5-10 minutes of warmup, followed by 3-4 multi-joint exercises for major muscle groups, comprising 2 sets of 10 to 25 repetitions at 40% of the one-repetition maximum (1-RM) for each exercise. Afterwards the aerobic part of the training will consist of 10-15 minutes of aerobic exercises (treadmill or outside walking or running, stationary cycling or outdoors or elliptical trainer) at 60-70% of peak VO2 or RPE 6-7 at Borg scale.
  The intensity will increase on weeks 9-26 after surgery to 4-5 multi-joint exercises of 3-4 sets of 10 to 25 repetitions and 30 minutes of aerobic exercises at 65-80% of peak VO2 or RPE 6-8 at Borg scale.
  Interventions: Other: Physical activity training
- The control group (No Intervention): The control group will receive routine health care without exercise supervision (clinical and nutritional follow up).

INTERVENTIONS:
Other: Physical activity training — Participants will be randomized into either one of three intervention groups (aerobic training, resistance training, or combined training comprised of resistance and aerobic training) and a control group. Training is described in the arm description section.
  Arms: Aerobic exercise training; Combination exercise training; Resistance exercise training

SUMMARY:
This study aims to determine how different types of exercise regimens (resistance, aerobic, or combined exercise regimens) can be used to minimize muscle loss and mobilize body fat in severely obese patients after bariatric surgery (BS), despite the rapid surgery-induced weight loss. Additionally, the study will examine how changes in the intestinal microbiota following BS act as a mediation factor that alter tissue-specific responses in muscle and adipose tissue. The study will also evaluate the effect of different types of exercise regimens on cardiometabolic markers, endocrine response, and physical function following BS.

Sixty sedentary (regular exercise <1 hour per week) candidates to bariatric surgery at Herzliya Medical Center will be recruited to participate in this six-month-long randomized control study. Participants will be randomly assigned to either one of three exercise regimens intervention groups (aerobic, resistance, or a combined exercise regimen combining aerobic and resistance exercises) or a control group that will receive standard care. Training will be supervised and matched for metabolic equivalent (METs). The intervention will take place at the Sylvan Adams Sports Institute at Tel Aviv University and an online platform.

All measurements will be taken at a presurgical baseline assessment and throughout the study, and will include changes of muscle mass and adipose tissue distribution, measured by a 3-Tesla magnetic resonance imaging (MRI); body composition- will be assessed using multichannel bioelectrical impedance (Seca); Bone mass, will be measured by a Dual-energy X-ray absorptiometry (DEXA); microbiota composition and changes will be evaluated by stool samples that will be subjected to 16S ribosomal ribonucleic acid (16s rRNA) profiling and metagenomics analysis; fasting blood samples will be used to examine endocrine control and cardiometabolic markers; anthropometric measurements to assess surgery results associations with physical activity outcomes and physical function will be assessed by several validated performance assessments, including handgrip, six-minute walk, sit-to-stand, maximum voluntary contraction, and maximal oxygen consumption (VO2max).

DETAILED DESCRIPTION:
The primary aim will be to determine how different types of exercise regimens (resistance, aerobic, or combined exercise regimens) can be used to minimize muscle loss and mobilize body fat in severely obese patients after BS, despite the rapid surgery-induced weight loss.

Secondary aims will include: I. To examine the effect of different exercise regimens on the composition and diversity of microbiomes, and their role in mediating muscle mass preservation following BS. II.Evaluate changes in cardiometabolic markers and endocrine response to different exercise regimens and evaluates microbiome mediation of these changes after BS. III.Assess the effect of different exercise regimens on physical function among patients following BS. IV.Clarify the mechanisms of muscle preservation and fat loss involving hormonal response and atrophy related-genes expression.

After baseline measurements (detailed below), participants will be randomized into one of four groups: 1. control group (n=15) that includes routine health care; 2. aerobic exercise training group (n=15), 3. resistance exercise training group (n=15), 4. combined aerobic and resistance exercise training group (n=15). Training sessions will be both in-person and as online exercise supervision. All groups will be supported by a dietitian as part of the routine health care after the bariatric surgery. The dietetic program for all groups will consist of a balanced diet by diet progression guidelines for bariatric patients (XX,ZZ) and the bariatric food pyramid (55). The protein content will be a minimum of 60 gr/protein per day, according to current guidelines (XX,ZZ) . Each training session will increase gradually up to 60 minutes per session, three times a week. Participants will be randomized into 4 groups for 26 weeks of intervention including aerobic, resistance, combined exercise training (aerobic + resistance) and a control group without exercise training.

All exercise training will be matched in metabolic equivalent (METs) and the time of training per week. Participants will begin a two weeks exercise adaptation period at 3-4 postoperative weeks. The activity adaptation plan will consist of 15-20 min. of walking, three times per week, at an intensity of 40-60% of peak oxygen consumption (VO2) or rate of perceived exertion (RPE) 4-6 on the Borg scale for all intervention groups. Following this period, each group will participate in a specific progressive training with the following regimen:

1. Aerobic exercise training group, weeks 5-8 after surgery: this training will consist of 30 min. of walking, 3 times per week at an intensity of 60-70% of peak VO2 or RPE 6-7 on Borg scale.

   Weeks 9-26 after surgery: this training will consist of 60 minutes of exercise, 3 times per week at an intensity of 65-80% of peak VO2 or RPE 6-8 on the Borg scale. The aerobic exercises will consist of a treadmill or outside walking or running, stationary cycling or elliptical trainer in continuous and interval training.
2. Resistance exercise training group, weeks 5-8 after surgery: this training will consist of 5-10 minutes of warmup, followed by 6-8 multi-joint exercises for major muscle groups, comprising 2 sets of 10 to 25 repetitions at 40% of the one-repetition maximum (1-RM) for each exercise. The intensity will increase on weeks 9-26 after surgery to 8-10 multi-joint exercises of 3-4 sets of 10 to 25 repetitions. For this training participants will use free-weights and bodyweight exercises.
3. The combination exercise training will consist of a combined aerobic and resistance exercise training sessions three times weekly. At weeks 5-8 after surgery, the sessions will include 5-10 minutes of warmup, followed by 3-4 multi-joint exercises for major muscle groups, comprising 2 sets of 10 to 25 repetitions at 40% of the one-repetition maximum (1-RM) for each exercise. Afterward, the aerobic part of the training will consist of 10-15 minutes of aerobic exercises (treadmill or outside walking or running, stationary cycling or outdoors or elliptical trainer) at 60-70% of peak VO2 or RPE 6-7 at Borg scale.

   The intensity will increase on weeks 9-26 after surgery to 4-5 multi-joint exercises of 3-4 sets of 10 to 25 repetitions and 30 minutes of aerobic exercises at 65-80% of peak VO2 or RPE 6-8 at Borg scale.
4. The control group will receive conventional treatment so as the other groups (medical and nutritional follow up).

ELIGIBILITY:
Inclusion Criteria:

* Sedentary participants: regular exercise performed <1 hour per week
* Candidates for primary bariatric surgery at Herzliya Medical Center in accordance to the National Institutes of Health (NIH) criteria for surgery: (body mass index (BMI) > 40 without coexisting co-morbidities or BMI > 35 with > 1 severe obesity-related comorbidities)
* Sex: all
* Age: 18 to 65 years.

Exclusion Criteria:

* Severe cardiopulmonary disease (e.g., recent myocardial infarction or unstable angina)
* Musculoskeletal or neuromuscular impairments that preclude exercise training
* Cognitive impairments
* Use of drugs that affect bone or muscle metabolism (mainly steroids)
* Patients with previous bariatric surgery

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Muscle mass (cm3) | At baseline and after 26 weeks of intervention
  Changes in thigh muscles volume
Body composition - fat mass | At baseline and after 13 and 26 weeks of intervention
  Fat mass (Kg)
Body composition | At baseline and after 13 and 26 weeks of intervention
  Fat free mass (Kg)

SECONDARY OUTCOMES:
Microbial composition and changes | At baseline and after 13 and 26 weeks of intervention
  16S rRNA profiling
Blood measurements - cardiometabolic markers | At baseline and after 13 and 26 weeks of intervention
  Cardiometabolic markers: Glucose (mg/dl), lipid profile (total cholesterol in mg/dl, HDL in mg/dl, LDL in mg/dl)
Blood measurements - Insulin | At baseline and after 13 and 26 weeks of intervention
  Insulin (pmol/L)
Blood measurements for skeletal muscle metabolism assessment | At baseline and after 13 and 26 weeks of intervention
  Levels of anabolic hormones such as growth hormone (ng/ml) (GH), insulin like growth factor (ng/ml) (IGF-1).
  Marker of inhibition of skeletal muscle growth: Myostatin (ng/ml)
Blood measurements - Inflammatory markers | At baseline and after 13 and 26 weeks of intervention
  Interleukin-6 (pg/ml) (IL6)
Blood measurements for nutritional status | At baseline and after 13 and 26 weeks of intervention
  Markers for nutritional status: Hemoglobin (g/dl), albumin (g/dl)
Blood measurements for micronutrients | At baseline and after 13 and 26 weeks of intervention
  Ferritin (ng/ml), B12 (ng/ml)
Blood measurements for liver function | At baseline and after 13 and 26 weeks of intervention
  Liver enzymes: alanine aminotransferase in units per liter (U/L) (AST), gamma-glutamyltransferase (U/L)(GGT), alanine aminotransferase (U/L) (ALT), alkaline phosphatase (U/L) (ALP);
Blood measurements of adipokines - leptin | At baseline and after 13 and 26 weeks of intervention
  Leptin (ng/ml)
Blood measurements of adipokines - adiponectin | At baseline and after 13 and 26 weeks of intervention
  Adiponectin (μg/ml)
Blood measurements for bone status | At baseline and after 13 and 26 weeks of intervention
  Blood bone markers such as Collagen Type-1 C-Telopeptide in μg/L (CTX) and total procollagen type 1 N-terminal propeptide in μg/L (P1NP).
Bone density changes | At baseline and after 13 and 26 weeks of intervention
  Assessed by DEXA scan (T score and g/cm^2)
Anthropometric measurements - BMI | At baseline and after 13 and 26 weeks of intervention
  Weight (kg) and height (m) will be combined to calculate BMI (kg/m^2)
waist circumference as part of Anthropometric measurements | At baseline and after 13 and 26 weeks of intervention
  waist circumference (cm)
Weight loss percentage outcomes | At baseline and after 13 and 26 weeks of intervention
  % Excess weight loss (%EWL) will be calculated by [(initial weight (kg))-(post operative weight(kg))] / [(initial weight in kg) - (ideal body weight in kg)].
  Total weight loss % (TWL%) will be calculated by [(initial weight (kg))-(post operative weight(kg))] / initial weight (kg).
Resting metabolic rate | At baseline and after 13 and 26 weeks of intervention
  measurement of resting daily energy expenditure (Kcal) will be measured by indirect calorimetry (Kcal/day) and energy expenditure per body kilogram per day (Kcal/Kg/day).

OTHER OUTCOMES:
Quality of life (QoL) | At baseline and after 13 and 26 weeks of intervention
  Will be assessed by the Bariatric Analysis and Reporting Outcome System (BAROS) questionnaire- measured by the results score
Physical function - 6 min walk test | At baseline and after 13 and 26 weeks of intervention
  6 min walk test will be assessed in meters
Physical function - sit to stand test | At baseline and after 13 and 26 weeks of intervention
  Sit to stand test will be assessed in seconds
Strength assessment | At baseline and after 13 and 26 weeks of intervention
  Will be assessed by performance tests Handgrip test (kg), Estimated one-repetition maximum (the maximum weight a participant can lift, in one attempt, in the bench press and leg press in kg)
Nutritional intake | At baseline and after 13 and 26 weeks of intervention
  Will be assessed by validated questionnaires such as food diary. Macronutrients composition will be measured from the self-reported nutritional intake: kcal daily intake, protein intake (in gr and in %of total kcal), carbohydrate intake (in gr and in %of total kcal) and fat intake (in gr and in %of total kcal).
Aerobic fitness - Cardio pulmonary exercise testing | At baseline and after 13 and 26 weeks of intervention
  Measurement of submaximal aerobic capacity will be assessed by oxygen consumption (indirect calorimetry) performed on a cycling ergometer, with VO2 reported in ml/kg/min.

CONTACTS AND LOCATIONS:
Overall Officials: Yftach Gepner, Ph.D., Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Other, Israel

IPD SHARING:
Plan to Share IPD: No